CLINICAL TRIAL: NCT03089567
Title: Comparison of the Salivary Levels of Streptococcus Mutans in Pediatric Patients With Early Childhood Caries After the Application of Silver Diamine Fluoride or 5% Sodium Fluoride Varnish
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was not conducted. No participants were enrolled
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMAHEN
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries
Keywords: Silver diamine Fluoride; Streptococcus mutans; Caries prevention; Fluoride
MeSH Terms: conditions — Dental Caries | interventions — Sodium Fluoride; Duraflor; silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CONTROL GROUP (No Intervention): Patients waiting for treatment under general Anesthesia without any intervention
- Sodium Fluoride Varnish (Active Comparator): Sodium Fluoride Varnish will be applied at 0,1,3 months Follow ups while waiting to receive dental treatment under general anesthesia
  Interventions: Drug: Sodium Fluoride
- Silver Diamine Fluoride (Experimental): Silver Diamine Fluoride will be applied at 0,1,3 months Follow ups while waiting to receive dental treatment under general anesthesia
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Sodium Fluoride — 5% Sodium Fluoride Varnish used for dental caries prevention and desensitizer
  Other Names: Duraflor
  Arms: Sodium Fluoride Varnish
Drug: Silver diamine fluoride — 38% Silver Diamine Fluoride used for dental caries prevention and desensitizer
  Other Names: Advantage Arrest
  Arms: Silver Diamine Fluoride

SUMMARY:
Comparison of the salivary levels of Streptococcus mutans in pediatric patients with Early Childhood Caries after the application of Silver Diamine Fluoride or 5% Sodium Fluoride Varnish

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease in children (Benjamin, 2010). Studies suggest there is a positive correlation between bacterial titers of Streptococcus mutans and dental caries (Pannu et. al., 2013). National surveys suggest children 2 to 5 years old have 27.90% of primary teeth with caries. This number near doubles to 51.17% for children 6 to 11 years old (United States, National Health and Nutrition Examination Survey, 1999-2004). The American Academy of Pediatric Dentistry discusses this prevalence, in particular the finding of caries in young children, calling it early childhood caries (ECC), defined as "the presence of 1 or more decayed (noncavitated or cavitated lesions), missing (due to caries), or filled tooth surfaces in any primary tooth in a child 71 months of age or younger" or severe early childhood caries (S-ECC), defined as any sign of smooth surface caries in children younger than three years of age (AAPD, 2008). Oral health disparities also vary by race, ethnicity and socioeconomic status. Among children ages 3-5 years old, the prevalence of dental caries was significantly higher for non-Hispanic black individuals, 19%, compared to non-Hispanic white individuals, 11%. Furthermore, the prevalence of dental caries was nearly twice as high for Hispanic individuals, 26%, compared to non-Hispanic white individuals (Dye et. al., 2012).

The use of fluoride in dentistry has played a significant role in reducing the prevalence and severity of dental caries. Water fluoridation is considered to be one of the ten greatest achievements in public health of the twentieth century (CDC, 1999). Sodium Fluoride (SF) varnishes have become a mainstay in many pediatric dental practices. Despite their intended use as desensitizing agents, fluoride varnishes are used routinely to inhibit the demineralization of enamel, promote remineralization of enamel, and arrest early enamel carious lesions (Chu et. al, 2008, CDC 2001). Fluoride also interferes with cariogenic bacteria's ability to metabolize carbohydrates, reducing their acid production, and ability to adhere to tooth surfaces, possibly reducing their ability to initiate decay (CDC, 2001). The ability of fluoride, namely SF varnishes to effect bacterial counts of S. mutans has been described in a limited extent in the literature. Chandak describes fluoride varnish's ability to reduce S. mutans counts in dental plaque, suggesting another way fluoride aids in the reduction on dental caries (Chandak et. al., 2016). However, other studies do not support SF varnishes abilities to significantly reduce plaque S. mutans counts (Sajjan, et. al., 2013). Other studies attempt to examine the effects of fluoride varnishes' ability to effect S. mutans adherence and biofilm formation. In their study Chau et. al, described a reduction in S. mutans adhesion and subsequent biofilm accumulation in the presence of a number of commercially available SF varnishes (Chau et. al, 2014).

Similar to fluoride compounds, the antimicrobial effects of silver containing compounds have been used in dentistry for nearly a century. The mechanism behind these compounds' antibacterial effect is derived from the bioactive silver ion's ability to disrupt and irreversibly damage vital bacterial enzyme systems (Lansdown 2006). Despite their use internationally since the early twentieth century, silver containing compounds have fallen out of favor over time. More recently, silver diamine fluoride (SDF), currently approved by the FDA for treatment of dentinal hypersensitivity, has been shown to possess caries arresting properties. The clinical applications of SDF are seemly vast. Average operating room (OR) wait times vary between providers and can range from days to months depending on such factors as the provider's availability and resources, the patient's symptomatology, medical history, and extent of treatment. The patient population served at the Yale-New Haven Hospital Pediatric Dental Center is diverse both demographically and medically. Due to the demand and need for comprehensive dental treatment under general anesthesia, average OR wait times are 4 to 6 months. Indications for OR treatment include medically complex patients, uncooperative or pre-cooperative behavior profiles, patients with extensive and multi-quadrant decay patterns, and patients who do not meet selection criteria for sedation modalities. SDF's ability to arrest dental decay allows for patients on lengthy wait list awaiting treatment in the OR to avoid having their caries progress significantly. SDF is not a solution to caries; however it can be a useful tool in stemming the progression of decay for children awaiting surgical intervention under general anesthesia.

In light of SDF's ability to arrest dental caries, there is a question about its ability to impact the etiology of caries initiation, namely its effect on salivary S. mutans counts in the oral cavity. Few studies have investigated SDF's ability to alter bacterial counts in the oral environment in children. The application of SDF to human dentin blocks resulted in the development of fewer colony forming units of a number of cariogenic bacteria, including S. mutans, compared to the control group (Mei, 2013). Similar results were described in a study examining the effect of silver fluoride on S. mutans biofilm formation (Knight et. al., 2009). The impact of such an effect would be profound and could change caries management and prevention in the pediatric population (Duangthip, Chu et. al. 2016).

The increased interest and popularity of SDF has the potential to change the manner in which dental caries are treated in the pediatric population. Applications can prevent more invasive and costly need for general anesthesia, or other advanced behavior management techniques, or possibly prevent the progression of decay and avoid the loss of teeth (Chu, 2000). Furthermore, the potential ability of SDF to affect the bacterial composition of the oral environment, possibly reducing the initiation of caries has the exciting potential to be a ground breaking public health achievement.

Hypothesis

Application of SDF on carious teeth will show a higher decrease the salivary bacterial counts of S. mutans form baseline in 2-6 years old patients with ECC when compared to S. mutans levels after sodium fluoride varnish application and no treatment

Preliminary Research Design

Patient selection: Healthy 2-6 years old patients with ECC awaiting comprehensive dental treatment under general anesthesia

Inclusion criteria: ASA I without prior history of dental restorations

Exclusion criteria: Patient with: special healthcare needs, xerostomia, complicated medical history (ASA II-VI)

Experimental Groups:

* 30 Patients that will receive 38% SDF application
* 30 Patients that will receive 5% NaF varnish application
* 30 Patient in Control group that will receive no treatment

Salivary collection: Salivary samples will be collected with SalivaBio Children's Swab.

A baseline S. mutans level will be obtained and quantified using Saliva-Check Mutans (GC America).

All carious teeth will receive a rubber cup and paste dental prophylaxis followed by either a topical application of 38% SDF, or 5% NaF varnish or no topical treatment.

Follow up: Further measurement of S. mutans levels will be obtained at 1, 3, 6 months after initial SDF, NaF varnish applications no treatment, without dental prophylaxis. Following salivary sample collections, re-application of SDF and NaF varnish will be applied to appropriate patient groups, and no further treatment provided to control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I without prior history of dental restorations

Exclusion Criteria:

* Patient with: special healthcare needs, xerostomia, complicated medical history (ASA II-VI)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Salivary levels of Streptococcus mutans | Baseline
  Salivary samples will be obtained with Children's Swab (SalivaBio) and S. Mutans level will be measured using Saliva-Check Mutans (GC America)
Salivary levels of Streptococcus mutans | 1 month
  Salivary samples will be obtained with Children's Swab (SalivaBio) and S. Mutans level will be measured using Saliva-Check Mutans (GC America)
Salivary levels of Streptococcus mutans | 3 months
  Salivary samples will be obtained with Children's Swab (SalivaBio) and S. Mutans level will be measured using Saliva-Check Mutans (GC America)
Salivary levels of Streptococcus mutans | 6 months
  Salivary samples will be obtained with Children's Swab (SalivaBio) and S. Mutans level will be measured using Saliva-Check Mutans (GC America)

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Lee, DMD, Principal Investigator — Yale New Haven Hospital; Christel Haberland, DDS, Principal Investigator — Yale New Haven Hospital

IPD SHARING:
Plan to Share IPD: Undecided